CLINICAL TRIAL: NCT04360772
Title: Monitoring of Corticosteroids Induced Immunosuppression Using mHLA-DR
Brief Title: Monitoring of Corticosteroids Induced Immunosuppression Using Monocyte Human Leukocyte Antigen-DR (mHLA-DR).
Acronym: HLA-DR
Status: Withdrawn | Type: Observational
Why Stopped: project cancelled
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL19_1029
Record Dates: First submitted 2020-04-15; First posted 2020-04-24 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Immunosuppression
Keywords: any pathology; corticosteroids therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: mHLA-DR — * Before treatment/ At inclusion/Day 0 : Collection of gender, date of birth, comorbidities, pathology implicating treatment by corticosteroids and other treatment administered at the time of inclusion.
  * At Day 0, Month 1, Month 3, Month 6 : Blood sampling (3mL) to proceed to mHLA-DR measurement. At those time-points, results from lymphocytes immunophenotyping, C-reactive protein and numeration will be collected.
  * At Month 24 : Collection from medical report of
  * any infectious events that would have occured during the follow-up
  * course of the disease with corticosteroids
  * survival or death at 24 months of follow-up.

SUMMARY:
Corticotherapy is widely used in auto-immune diseases. If induced immunosuppression by corticosteroids is well admitted, it's currently not possible to determine individual risk of infection. Thus, the development of new biomarkers able to reflect immunological status under immunosuppressive treatments is needed. It would help identifying patients who would benefit from adapted treatment protocols or infectious prophylaxis. In this field, the mHLA-DR (monocyte Human Leukocyte Antigen-DR) has shown encouraging results. However, it has never been used in patients treated by immunosuppressive therapies. The investigators aim to describe changes induced by corticosteroids in mHLA-DR expression in vivo. To achieve this goal, the investigators will measure mHLA-DR before treatment, after 1 months, 3 months and 6 months of treatment. Finally, the investigators will look for correlation between the level of expression of mHLA-DR and the cumulated dose of corticosteroids administered.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged of 18 years old or more, male or female.
* Patient diagnosed with any pathology indicating a treatment by corticotherapy at 1mg/kg/day.
* Patient who didn't express any opposition to be enrolled in the study after reading the dedicated information letter.
* Patient affiliated to social heath care regimen

Exclusion Criteria:

* Treatment by corticosteroids in the previous 6 months.

  * Immunsuppressive treatment (except for corticosteroids) in the previous 2 years.
  * Patient under judicial protection, guardianship or curators

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient Diagnosed With Any Pathology Indicating a Treatment by Corticotherapy
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Kinetics of mHLA-DR expression determined by flow cytometry before treatment and during the 6 first months of degressive corticosteroids doses | Month 1, 3 and 6
  mHLA-DR expression level will be compared between :
  * Before treatment and at 1 month of treatment
  * Before treatment and at 3 months of treatment
  * Before treatment and at 6 months of treatment
  * 1 month and 3 months of treatment
  * 1 month and 6 months of treatment

CONTACTS AND LOCATIONS:
Overall Officials: ARNAUD HOT, MD, Principal Investigator — Service de Médecine Interne